CLINICAL TRIAL: NCT04905121
Title: An Exploratory Open-Label, Phase 1b, Ascending Dose Study to Evaluate the Effects of Oral 3-[2-(Dimethylamino)Ethyl]-1h-indol-4-yl Dihydrogen Phosphate (Psilocybin, BPL-PSILO) on Cognition in Patients With Chronic Short-Lasting Unilateral Neuralgiform Headache Attacks (SUNHA)
Brief Title: Phase 1b Study in Patients With Short-Lasting Unilateral Neuralgiform Headache Attacks (SUNHA)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit patient population
Sponsor: Beckley Psytech Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPL-PSILO-101
Record Dates: First submitted 2021-05-06; First posted 2021-05-27 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Short Lasting Unilateral Neuralgiform Headache Attacks
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: An exploratory open-label phase 1b, ascending dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin will be provided in form of dry filled capsules and administered orally in three ascending doses

SUMMARY:
This exploratory open-label phase 1b, ascending dose study is to evaluate the effects of psilocybin on cognition in patients with Chronic Short-Lasting Unilateral Neuralgiform Headache Attacks (SUNHA)

DETAILED DESCRIPTION:
The study aims to:

Determine the safety and tolerability of psilocybin when administered to patients with chronic SUNHA

Determine the effects of psilocybin on cognition when administered to patients with chronic SUNHA

Explore the change in frequency, duration, and intensity of headache attacks with escalating doses of psilocybin in patients with chronic SUNHA

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic SUNHA

Exclusion Criteria:

* Other comorbidities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with treatment emergent AEs (TEAES) | From first dose administered through to the last follow up visit, approximately 39 days
Treatment-related changes in Paired Associates Learning (PAL) scores and evaluation of dose response | From first dose administered until the las dose administered, approximately 11 days
Treatment-related changes in Spatial Working Memory (SWM) scores and evaluation of dose response | From first dose administered until the las dose administered, approximately 11 days
Treatment-related changes in Reaction Time Index (RTI) scores and evaluation of dose response | From first dose administered until the las dose administered, approximately 11 days
Treatment-related changes in Rapid Visual Information Processing (RVP) scores and evaluation of dose response | From first dose administered until the las dose administered, approximately 11 days
Change in frequency of headache attacks | From screening until the follow up visit, approximately 39 days
Change in duration of headache attacks | From screening until the follow up visit, approximately 39 days
Change in intensity of headache attacks | From screening until the follow up visit, approximately 39 days
  Patients will complete a diary on a daily basis and capture the intensity of their headaches by assigning a score out of 10 where 0 is pain free and 10 is excruciating pain

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the UK GDPR, individual participant data will not be shared publicly. Group data will be presented in publication after study completion.